CLINICAL TRIAL: NCT01386697
Title: A Prospective Radiation Oncology Planning Study For Lung, Gastrointestinal And Lymphomatous Malignancies Using Proton Radiotherapy As Compared To 3D Conformal And Intensity-Modulated X-Ray Therapy For Dosimetric Evaluation Of Tumoral Coverage And Dose To Organs-At-Risk.
Brief Title: DIBH Proton Planning
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 13910
Record Dates: First submitted 2011-06-30; First posted 2011-07-01 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Lung Cancer; Breast Cancer; Gastrointestinal; Lymphomatous Malignancies
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The overall objective is to estimate the actual or potential benefit of deep inspiration breath holding (DIBH) treatment in the context of proton radiotherapy as compared to 3 dimensional conformal radiation therapy (3DCRT) and intensity-modulated x-ray therapy (IMXT), as it relates to variability in tumor localization, treatment margins, target volume definition, doses to organs at risk and variations with treatment planning.

DETAILED DESCRIPTION:
Image acquisition and treatment under deep inspiration breath hold (DIBH) has been demonstrated to reduce treated volumes and doses to organs at risk (OARs) for photon radiotherapy but has not been investigated in the context of proton radiotherapy. The objective of this registry study is to prospectively evaluate deep inspiration breath hold CT scans for use in proton radiotherapy treatment planning and obtain dosimetric data to assess for changes in target volume, planning volumes and doses both to tumor and organs at risk using the SpiroDynrX (SDX) deep inspiration breath hold system as compared to free breathing and 4D CT scans. Patients will be treated with photon therapy. This is a prospective non-randomized, single arm, single institution registry study of patients undergoing definitive external beam photon radiotherapy in our department. Deep inspiration breath hold CT scans will be obtained in our department in the treatment position at the time of CT simulationin addition to the currently obtained free breathing and 4D CT scans. These scans will all be co-registered with the treatment planning CT. Treatment planning volumes will be delineated by the physician and compared to the results and data for our current standard of care utilizing 4D CT scans. Patients will be treated with breath hold CT using photon radiotherapy but we will prospectively create proton treatment plans which will also be compared to the photon treatment plans used for actual treatment. Variability in tumor localization, target volume definition, doses to organs at risk and treatment planning particularities will be summarized and reported across several modalities, including: 3 dimensional conformal radiation therapy (3DCRT), intensity-modulated x-ray therapy (IMXT) and proton therapy. Correlations will be statistically analyzed and reported in terms of minimum, maximum, average and standard deviation, and other dose volume histogram parameters, and where appropriate, compared with appropriate statistical methods (for example, student t-test).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Biopsy-proven malignancy
* The diagnosis of hepatocellular carcinoma may be made on a clinical basis without the need for a biopsy if the following criteria are met: a) Documentation of hepatitis B or C infection b)Liver mass with characteristic imaging (CT or MRI) features of hepatocellular carcinoma c) Alpha-feta protein (AFP) level greater than 20 ng/mL 3. Planned curative external beam RT as part of the patients treatment for the cancer diagnosis.
* Subject must be cable of giving informed consent for standard external beam radiation therapy as well as for the study.
* Subjects must be able to tolerate the deep inspiration breath hold (DIBH) training and procedures.

Exclusion Criteria:

* Subjects unsuitable for or unable to undergo definitive external beam, radiation therapy for their diagnosis of cancer
* Subjects undergoing radiation with palliative (i.e., non-curative) intent.
* Subjects unwilling to undergo simulation with the SpiroDynrX (SDX) system.
* Subjects unable to hold their breath for a minimum of 10 seconds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This registry study will enroll patients who are 18 years of age or older who select to undergo external beam radiation therapy as definitive or adjuvant treatment for their diagnosis of lung, breast, gastropintestinal or lymphomatous malignancies in the Department of Radiation Oncology.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Plastaras, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States